CLINICAL TRIAL: NCT07080268
Title: Validation of a Questionnaire for Quality of Life Assessment in Patients With Transthyretin Amyloidosis in Argentina.
Brief Title: Validation of a Questionnaire for Quality of Life Assessment in Patients With Transthyretin Amyloidosis.
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Principal Investigator, Fernando Torres, PhD, Hospital General de Niños Pedro de Elizalde
Other Study IDs: HGNPE
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Amyloidosis in Transthyretin (TTR); Hereditary Amyloidosis, Transthyretin-Related
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic patients with hereditary amyloidosis

SUMMARY:
Prospective study of development and validation of a questionnaire on quality of life in patients with Hereditary Amyloidosis The questionnaire development process will include 4 medical specialists experts in Transthyretin Amyloidosis (2 neurologists, 1 cardiologist, 1 physician clinical/hepathologist), 1 psychologist; 1 social worker; and 3 patients (with confirmed Hereditary amyloidosis) members of ALAPA. (Local PAG)

Population and sample:

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed ATTR (genetic test), older than 18 years old in stage I, II and III of the PND scale (polyneuropathy disability: I Sensory neuropathy ; II Motor symptoms, but with preserved ambulation; IIIa Requires 1 cane to ambulate; IIIb requires two canes/walker).

Exclusion Criteria:

* patients who participated in the validation process of the questionnaire: patients who participated in the questionnaire construction process or adjustments to the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed ATTR (genetic test), older than 18 years in stage I, II and III of the PND (polyneuropathy disability) scale
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To develop and validate a structured and self-administered quality of life questionnaire in patients with hereditary amyloidosis | 6 months
  To develop and validate a structured and self-administered questionnaire specific to covering physical, emotional and social aspects, to assess the impact of hereditary transthyretin amyloidosis on the quality of life of patients residing in Argentina.

CONTACTS AND LOCATIONS:
Locations (1):
- HGNPE, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conceicao I, Coelho T, Rapezzi C, Parman Y, Obici L, Galan L, Rousseau A. Assessment of patients with hereditary transthyretin amyloidosis - understanding the impact of management and disease progression. Amyloid. 2019 Sep;26(3):103-111. doi: 10.1080/13506129.2019.1627312. Epub 2019 Jul 24. PMID 31339362
- [Background] Aimo A, Rapezzi C, Perfetto F, Cappelli F, Palladini G, Obici L, Merlini G, Di Bella G, Serenelli M, Zampieri M, Milani P, Licordari R, Teresi L, Ribarich N, Castiglione V, Quattrone F, De Rosis S, Vergaro G, Panichella G, Emdin M, Passino C. Quality of life assessment in amyloid transthyretin (ATTR) amyloidosis. Eur J Clin Invest. 2021 Nov;51(11):e13598. doi: 10.1111/eci.13598. Epub 2021 May 22. PMID 33982288